CLINICAL TRIAL: NCT01916018
Title: Phenotype and Genotype Analysis in Congenital Hypothyroidism Due to Thyroid Dysgenesis. The Use of Genetic Analysis in the Early Care of Children With Thyroid Dysgenesis
Brief Title: Clinical and Genetic Analysis in Congenital Hypothyroidism Due to Thyroid Dysgenesis.
Acronym: HYPOTYGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P11012-IDRCB 2012-A00797-36
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Congenital Hypothyroidism
Keywords: Congenital hypothyroidism; Thyroid dysgenesis; Genetics; Associated malformations; Psychomotor delay; Mental retardation
MeSH Terms: conditions — Congenital Hypothyroidism; Thyroid Dysgenesis; Learning Disabilities; Intellectual Disability | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hypothyroid group (Other): Clinical exams radiologic exams Blood sample
  Interventions: Other: Clinical and radiologic exams and blood samples

INTERVENTIONS:
Other: Clinical and radiologic exams and blood samples

SUMMARY:
Congenital hypothyroidism (CH) is a rare disease that affects 1 in 3500 newborn. This condition is detected consistently since the late 1970s in France, which has led to early care and a significant improvement in prognosis and intellectual stature of these children. However neurodevelopmental disorders persist in 10-15% of cases. More associated diseases have been reported in approximately 10% of cases. These observations are in most cases poorly understood. The family nature of the CH is now well recognized and a dozen genes involved up to now. However, in the majority of cases (HC not due to a disorder of the organification of iodine), few mutations have been found in the reported number of patients (5-10%), suggesting the involvement of other genes. Some of the genes have been implicated in particular specific syndromic forms but many pathological associations remain unexplained. Also, a more complete genetic elucidation of CH would enable a better understanding of its etiology and thus its risk of familial recurrence (frequently asked questions by parents of children with CH) and secondly the presence of associated pathologies.

Main goal: to describe the population with CH (not due to a disorder of the organification of iodine) not only on clinical, biological and radiological (phenotypic analysis) but also on the genetic level to establish a genotype / phenotype correlation.

DETAILED DESCRIPTION:
Congenital hypothyroidism (CH) is a rare disease that affects 1 in 3500 newborn. This condition is detected consistently since the late 1970s in France, which has enabled early care and a significant improvement of the intellectual stature and prognosis of these children. However neurodevelopmental disorders persist in 10-15% of cases. More associated pathologies have been reported in nearly 10% of cases. These observations are in most cases poorly understood. The family nature of the HC is now well accepted and a dozen genes is now involved. However in the majority of cases (HC not due to a disorder of the organification of iodine), few mutations have been found relative to the number of patients (5-10%), suggesting the involvement of other genes. Some of the genes have been implicated in such specific syndromic forms but many pathological associations remain unexplained. Also, a more complete elucidation of genetic HC enable a better understanding of its etiology and thus share the risk of familial recurrence (frequently asked by parents of children with questions) and secondly the presence of comorbidities.

Main objective: To describe the population with HC (not due to a disorder of the organification of iodine) not only on clinical, biological and radiological (phenotypic analysis) but also at the genetic level to establish a genotype / phenotype correlation.

Secondary objectives:

1. study the frequency of malformations and / or pathological associations in patients with HC
2. identify groups of patients with syndromic forms in whom early treatment may improve the prognosis of children
3. to search for mutations in genes known to be involved in the pathology
4. to search for new loci and / or genes involved
5. to determine the optimal genetic strategy to adopt before a HC case.

Inclusion criteria:

- Patient: Newborn (0-27 days) or infant (28 days-23 months), or a child or adult with congenital hypothyroidism (that is to say with a filter paper TSH > 15 mU / ml and / or a serum TSH> 10 mU / ml) diagnosed in the first months of life, regardless of age, sex, weight and size.

Subjects with blood levels of free thyroid hormones (FT3 and FT4) in the standards are described as having subclinical hypothyroidism.

If treatment with L-thyroxine has been stopped without relapse (that is to say, always with a TSH <5 mU / ml with different controls), hypothyroidism is called transient, whatever the age of discontinuation.

* No earlier or neonatal goitre by palpation or ultrasound examinations
* negative perchlorate test (ie rate of iodine salting <10% at 2 hours from the injection of the perchlorate) when the thyroid gland in place
* No self-immunity against thyroid in children and / or in her mother (defined by a antithyroperoxidase presence of antibodies and / or thyroglobulin)
* Signature of free and informed consent by the patient or his legal representative
* Affiliate or enjoying a social security system

Non-inclusion criteria:

* Presence of antithyroid autoimmunity in children and / or mother markers (antithyroperoxidase presence of antibodies and / or thyroglobulin)
* Goiter by neonatal palpation or ultrasound examinations
* positive perchlorate test (ie. decreased rate of iodine> 10% at 2 injection of perchlorate)

Exclusion criteria:

Patients of foreign origin returned to their country will be excluded from the study, even those who are lost to follow or refuse to perform additional tests requested.

* Acts / medical examinations carried out in taking care of but usually within the scope of the search if not done in the care:
* Ultrasound thyroid
* Thyroid scintigraphy
* Data on thyroid function: minimum values of FT3, FT4 and TSH plasma last blood test and current treatment (dose of L-T4)
* Data on the current education (or occupation) and level of psychomotor development established by the scale of Denver
* Data associated diseases: echocardiography and / or existence of heart disease and kidney and / or ultrasound existence of renal disease
* Clinical examination performed by the clinician investigator geneticist center.
* Standard karyotype
* Specific Genetic Analysis: TTF1/Nkx2.1; FOXE/TTF2; PAX8, TSHR and Nkx2.5 on blood sample for all patients (10 ml EDTA blood)
* Search for new genes

  1. cases of consanguineous families, a genome-wide study will be looking for homozygous regions shared by affected members (or homozygosity mapping autozygotie mapping).

     (in related first degree blood sample of 10 mL EDTA)
  2. for patients with one or more diseases associated with HC, seeking a number variation (CNV) of a gene or locus.

If abnormality found in the patient, blood samples of two parents 10 ml EDTA search CNV variation to exclude inherited CNVs.

350 patients with HC followed by endocrinologists and / or French pediatricians. Note that a majority of patients has been identified in the database of more than 10 years in the INSERM U845 (Necker Hospital, Paris).

Planned duration of the test: 42 month Time inclusions: 18 months Duration of follow-up: 2 years The patient may be contacted with the agreement at any time to perform additional tests required and / or a new blood sample for further genetic study.

Multinational cross-sectional study In a first period, it will accurately describe patients phenotypically and in a 2nd period, find a genetic cause. This will be facilitated by the presence of DNA already collected for the majority of them in one national bank in France, established in laboratory research center U845 (biocollection DC-2008-596, Faculty Necker, Paris)

Primary endpoint:

* Etiological type of congenital hypothyroidism: athyrose, ectopia, hemiagnÃ©sie, hypoplastic gland in place of normal shape and size
* Presence and type of cytogenetic abnormalities and / or genetically presence and type of pathology associated with HC
* Presence of neuropsychological abnormalities (including delayed psychomotor development)

Secondary endpoints:

Will be considered in this chapter all the elements that can cause psychomotor retardation (3):

* Time management of hypothyroidism
* Optimization of the treatment of hypothyroidism: delay normalization of TSH and T4, number of TSH> 15 mU / ml during follow-up, adherence
* The presence of an earlier complication and / or neonatal

Statistical analysis will include the following main chapters:

* Description of the population (anamnestic data, clinical, hormonal status at diagnosis and at follow-up imaging data).
* Analysis of the determinants of psychomotor development (see criteria secondary outcome).
* Data from the genetic study (type of mutated gene and nature of the mutation or genetic location of a deletion or duplication) An analysis of the observed association between mutations and phenotypes of patients will be performed by the methods of comparison genotype frequencies in different groups of subjects (chi-square test or Pearson 2 if necessary by the Fisher exact test).

The hazard ratios associated with the risk of occurrence of each event will be estimated with confidence intervals at 95%. Comparisons of events between different mutations will be tested using the log-rank test. All tests will be bilateral and a value of p <0.05 is considered statistically significant.

After 42 month, the study will identify the responsible genes in a large proportion of patients with congenital hypothyroidism (excluding disorders organification of iodine), to establish a genotype-phenotype correlation and propose early genetic screening (through systematic newborn screening) to patients and their families. The study of the frequency of associated diseases and genetic elucidation will also provide recommendations for early treatment (possibly "preventive") from other later predictable and potentially negative repercussions associated with hypothyroidism

ELIGIBILITY:
Inclusion Criteria:

- Patient: newborn (0-27 days) or infant (28 days 23 months), or child or adult with congenital hypothyroidism (that is to say with a TSH > 15 mU / ml at screening on filter paper and / or plasma TSH> 10 mU / ml) diagnosed in the first months of life, whatever their age, sex, weight and size.

Subjects with blood levels of free thyroid hormones (FT3 and FT4) in the standards will be described as having subclinical hypothyroidism.

If treatment with L-thyroxine could be stopped without relapse (that is to say, always with a TSH <5 mU / ml with different controls), hypothyroidism is said to be transient, whatever the age of discontinuation of treatment.

* No pre or neonatal goitre by palpation or ultrasound thyroid
* negative perchlorate test (ie decreased rate of iodine captation <10% at 2h injection of perchlorate) when the thyroid gland in place
* No self-immunity known to thyroid in children with and / or his mother (defined by a antithyroperoxidase antibodies and / or antithyroglobulin)
* Signature of free and informed consent by the patient or his legal representative
* Affiliation or enjoying a social security system

Exclusion Criteria:

* Presence of markers antithyroid autoimmunity in children and / or mother (antithyroperoxidase antibodies and / or antithyroglobulin)
* Pre or neonatal goiter on palpation or ultrasound thyroid
* Test positive perchlorate (ie salting rate of iodine> 10% at 2 injection perchlorate)
* Patients of foreign origin returned to their country will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
etiological type of the congenital hypothyroidism | 2 years
  Etiological Type of the congenital hypothyroidism: athyreosis, ectopia, hémiagenesis, hypoplastic gland in place of normal shape and size
Presence and type of cytogenetic and / or genetic abnormality associated with HC | 2 years
Presence and type of pathology associated with HC | 2 years
Presence of abnormal neuropsychological (including delayed psychomotor development) | 2 years

SECONDARY OUTCOMES:
time to treatment of hypothyroidism | 2 years
  Optimization of the treatment of hypothyroidism: normalization period of TSH and T4, TSH number of> 15 mU / ml during follow-up, adherence
Presence of a prenatal and / or neonatal complication | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric endocrinology gynecology and diabetology, Hôpital Necker Enfants Malades, Assistance Publique - Hôpitaux de Paris , Université Paris Descartes, INSERM unit U 845, Paris, France

REFERENCES:
- [Background] Stoupa A, Adam F, Kariyawasam D, Strassel C, Gawade S, Szinnai G, Kauskot A, Lasne D, Janke C, Natarajan K, Schmitt A, Bole-Feysot C, Nitschke P, Leger J, Jabot-Hanin F, Tores F, Michel A, Munnich A, Besmond C, Scharfmann R, Lanza F, Borgel D, Polak M, Carre A. TUBB1 mutations cause thyroid dysgenesis associated with abnormal platelet physiology. EMBO Mol Med. 2018 Dec;10(12):e9569. doi: 10.15252/emmm.201809569. PMID 30446499
- [Background] Carre A, Stoupa A, Kariyawasam D, Gueriouz M, Ramond C, Monus T, Leger J, Gaujoux S, Sebag F, Glaser N, Zenaty D, Nitschke P, Bole-Feysot C, Hubert L, Lyonnet S, Scharfmann R, Munnich A, Besmond C, Taylor W, Polak M. Mutations in BOREALIN cause thyroid dysgenesis. Hum Mol Genet. 2017 Feb 1;26(3):599-610. doi: 10.1093/hmg/ddw419. PMID 28025328
- [Derived] Stoupa A, Kariyawasam D, Nguyen Quoc A, Polak M, Carre A. Approach to the Patient With Congenital Hypothyroidism. J Clin Endocrinol Metab. 2022 Nov 25;107(12):3418-3427. doi: 10.1210/clinem/dgac534. PMID 36107810